CLINICAL TRIAL: NCT00002794
Title: Evaluation of Chemotherapy as Initial Treatment for Retinoblastoma
Brief Title: Carboplatin Plus Vincristine in Treating Children With Retinoblastoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000064874; P30CA021765 (NIH); P01CA023099 (NIH); SJCRH: RET3; NCI-H96-0935
Record Dates: First submitted 1999-11-01; First posted 2004-04-26 (Estimated); Last update posted 2011-10-04 (Estimated); Status verified 2011-10

CONDITIONS: Retinoblastoma
Keywords: intraocular retinoblastoma
MeSH Terms: conditions — Retinoblastoma | interventions — Carboplatin; Vincristine

INTERVENTIONS:
Drug: carboplatin
Drug: vincristine sulfate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of carboplatin plus vincristine in treating children with retinoblastoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Estimate the objective response rate in infants and children with retinoblastoma when treated with carboplatin (CBDCA) and vincristine (VCR) every 3 weeks for 24 weeks. II. Assess the success of this regimen in delaying radiotherapy and eliminating the need for surgery by estimating the cumulative incidence function of treatment failure. III. Estimate the cumulative incidence of failure of this regimen as measured by subsequent treatment with radiotherapy or surgery.

OUTLINE: All patients receive carboplatin and vincristine every 3 weeks for a maximum of 8 courses. Patients with disease progression after at least 2 courses are removed from study and considered for alternative therapy. Patients are followed every 6 weeks for 1 year, every 2 months for 1 year, every 3-4 months for 3 years, and yearly for 12 years.

PROJECTED ACCRUAL: A total of 25 patients will be accrued for this study within 4.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Newly diagnosed retinoblastoma Bilateral or multifocal unilateral disease in children under age 10 Unilateral, multifocal tumors less than 5 dd in children under age 2 No metastatic disease Disease evidenced by ophthalmoscopic/imaging exam, ultrasound, CT, or MRI Fundus drawings and photographs required

PATIENT CHARACTERISTICS: Age: 10 and under Performance status: Not specified Life Expectancy: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy Endocrine therapy: Not specified Radiotherapy: No prior radiotherapy Surgery: Not specified

Max Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 1996-02; Primary Completion 2001-06 (Actual); Study Completion 2001-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Rodriguez-Galindo, MD, Study Chair — St. Jude Children's Research Hospital
Locations (2):
- United States (2):
  - University of Tennessee, Memphis Cancer Center, Memphis, Tennessee
  - Saint Jude Children's Research Hospital, Memphis, Tennessee

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org